CLINICAL TRIAL: NCT03137277
Title: A Randomized Comparative Study Between Two Instrument Generations to Improve Adenoma Detection in Screening Colonoscopy
Brief Title: A Study Between Two Instrument Generations to Improve Adenoma Detection in Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Clinic Director of Interdisciplinary Endoscopy Department and Clinic, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV4343
Record Dates: First submitted 2017-04-19; First posted 2017-05-02 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Adenoma Detection Rate
Keywords: Colonoscopy; ADR; Adenoma detection rate; colonoscopic imaging feature improvement; Olympus colonoscopes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon Polyps and Adenoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Olympus 190: Olympus colonoscope 190 C (intervention group), screening colonoscopy examination with the latest generation colonoscope (190 series CF or PCF colonoscopies, Olympus Corp, Hamburg, Germany).
  Interventions: Procedure: screening colonoscopy
- Olympus 160/165: Olympus colonoscope 165 C (control group), screening colonoscopy examination with the 160/5 generation colonoscope (Olympus Corp, Hamburg, Germany),
  Interventions: Procedure: screening colonoscopy

INTERVENTIONS:
Procedure: screening colonoscopy — Introduction and forwarding of the device up to caecum/terminal ileum. Then withdrawal and inspection of colonic wall. Biopsies and polypectomies if necessary. overall and diagnostic (only withdrawal) times being recorded separately.
  Polyps are documented with regards to location (caecum, ascending, transverse and descending colon, sigmoid and rectum), size (open forceps or snare for comparison) and morphology using the Paris classification (polypoid pedunculated or sessile, non-polypoid slightly elevated/flat/depressed, ulcerous) Polyps were then resected using biopsy forceps or cold snare (for polyps < 5 mm), or conventional polypectomy according to local standards.

SUMMARY:
Adenoma detection rate (ADR) is the most important parameter to measure outcome quality of (screening) colonoscopy. Since single improvements of imaging have not been able to improve ADR in many randomized studies, the present study tested the hypothesis that only multiple imaging improvements such as seen with two generation changes of colonoscopies - i.e. skipping one colonoscope generation - may be necessary before improvements in ADR can be measured.

The investigators will test this hypothesis in the present randomized tandem study in 7 private practices in Hamburg and Berlin, in a pure screening colonoscopy setting, aiming at inclusion of 1200 patients > age of 55 years (screening colonoscopy cut-off in Germany). Exclusion criteria are symptomatic patients and colonoscopies planned for therapeutic reasons. Main outcome parameter is the ADR (rate of patients with at least one adenoma/all patients).

DETAILED DESCRIPTION:
The study was a prospective multicenter randomized study involving 7 private practice gastroenterology offices with a total of 14 experienced examiners (> 2000 colonoscopies), performed between November 2013 and September 2016 (sets of instruments were made available to 3-4 centers each during 6-12 months).Study population:

Patients were selected from the screening colonoscopy list (age ≥ 55 years), with further inclusion criteria being status 1 and 2 of the ASA classification. After informed consent, patients were randomized using sealed envelopes per center to one of either of the two study groups

1. 190 C group (intervention group), examination with the latest generation colonoscope (190 series CF or PCF colonoscopies, Olympus Corp, Hamburg, Germany).
2. 165 C group (control group), examination with the 160/5 generation colonoscope (Olympus Corp, Hamburg, Germany), Each patient underwent bowel preparation in accordance with local practice of the centers. Bowel cleansing quality was segmentally assessed using a modified overall "Boston Bowel Preparation Scale". Introduction and withdrawal times were measured, and times required for biopsies and polypectomies were considered separately, i.e. overall and diagnostic only withdrawal times were recorded separately.

Polyps were documented with regards to location (caecum, ascending, transverse and descending colon, sigmoid and rectum), size and morphology using the Paris classification (polypoid pedunculated or sessile, non-polypoid slightly elevated/flat/depressed, ulcerous). Polyps were then resected using biopsy forceps or cold snare or conventional polypectomy according to local standards. Histology of resected polyps was analyzed by local private practice specialized GI pathologists according to the Vienna classification with regards to dysplasia grade and the presence of serrated adenomas; final histologic categories were hyperplastic, adenomatous [tubulous, villous, tubulovillous, serrated (traditional or sessile serrated)]. Small distal rectal polyps were not systematically biopsied or resected, due to a very high likelihood to be hyperplastic.

ELIGIBILITY:
Inclusion Criteria:

* screening colonoscopy, age ≥ 55 years
* status 1 and 2 of the ASA classification
* signed informed consent

Exclusion Criteria:

* Symptoms indicative of colorectal disease such as colonic bleeding, significant diarrhea, obstipation and change in bowel habits
* Known colonic disease for further evaluation (e.g. inflammatory bowel disease, polyps for resection)
* Surveillance after polypectomy or colon tumor surgery
* Anticoagulants preventing biopsy or polypectomy
* Poor general condition (ASA III or more)
* Incomplete colonoscopy planned

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 55 years and above, planned for a screening colonoscopy in one of the parttaking private practices.
Sampling Method: Probability Sample
Enrollment: 1221 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | day 1
  adenoma detection rate (ADR) of 190 colonoscopes in comparison to 160/5 colonoscopes at the patient level (% of patients with at least one adenoma).

SECONDARY OUTCOMES:
Adenoma rate | through study completion, an average of 6 months
  Adenoma rate calculated at the adenoma level (all adenomas/all patients) and as the number of adenomas per adenoma carrier.
Adenoma subgroups: size | through study completion, an average of 6 months
  Adenoma subgroups due to size (< 1 cm, > 1 cm)
Adenoma subgroups: form | through study completion, an average of 6 months
  Adenoma subgroups due to form (flat, sessile, pedunculated)
Adenoma subgroups: location | through study completion, an average of 6 months
  Adenoma subgroups due to location (right sided - down to left hepatic flexure, left sided - descending colon, sigmoid and rectum)
Adenoma subgroups: histology | through study completion, an average of 6 months
  Adenoma subgroups due to histologic subgroups (SSA, HGIN)
Cecal intubation rate | through study completion, an average of 6 months
  Cecal intubation rate per arm, all patients
complication rate | through study completion, an average of 6 months
  Complications in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — University Hospital
Locations (7):
- Germany (7):
  - Gemeinschaftspraxis Hohenzollerndamm, Berlin
  - Gastroenterologie am Bayerischen Platz, Berlin
  - Praxis Mayr / Heller, Berlin
  - Dr. Alireza Aminalai, Berlin
  - Dr. Jens Aschenbeck, Berlin
  - Gastropraxis Eppendorferbaum, Hamburg
  - Gastroenterologie-Fontanay, Hamburg

IPD SHARING:
Plan to Share IPD: No
no individual participant data sharing

REFERENCES:
- [Background] Imperiale TF, Glowinski EA, Lin-Cooper C, Larkin GN, Rogge JD, Ransohoff DF. Five-year risk of colorectal neoplasia after negative screening colonoscopy. N Engl J Med. 2008 Sep 18;359(12):1218-24. doi: 10.1056/NEJMoa0803597. PMID 18799558
- [Background] Winawer SJ, Zauber AG, Gerdes H, O'Brien MJ, Gottlieb LS, Sternberg SS, Bond JH, Waye JD, Schapiro M, Panish JF, et al. Risk of colorectal cancer in the families of patients with adenomatous polyps. National Polyp Study Workgroup. N Engl J Med. 1996 Jan 11;334(2):82-7. doi: 10.1056/NEJM199601113340204. PMID 8531963
- [Background] von Karsa L, Patnick J, Segnan N. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Executive summary. Endoscopy. 2012 Sep;44 Suppl 3:SE1-8. doi: 10.1055/s-0032-1309822. Epub 2012 Sep 25. PMID 23012113
- [Background] Millan MS, Gross P, Manilich E, Church JM. Adenoma detection rate: the real indicator of quality in colonoscopy. Dis Colon Rectum. 2008 Aug;51(8):1217-20. doi: 10.1007/s10350-008-9315-3. Epub 2008 May 24. PMID 18500502
- [Background] Bretagne JF, Ponchon T. Do we need to embrace adenoma detection rate as the main quality control parameter during colonoscopy? Endoscopy. 2008 Jun;40(6):523-8. doi: 10.1055/s-2007-995786. Epub 2008 May 8. No abstract available. PMID 18464196
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Barclay RL, Vicari JJ, Doughty AS, Johanson JF, Greenlaw RL. Colonoscopic withdrawal times and adenoma detection during screening colonoscopy. N Engl J Med. 2006 Dec 14;355(24):2533-41. doi: 10.1056/NEJMoa055498. PMID 17167136
- [Background] Bock, J., Toutenburg, H. (1991). Sample size determination in clinical research. In: Rao, C.R., Chakraborty, R. (eds.): Handbook of statistics, Elsevier, 515 - 538.
- [Background] Adler A, Wegscheider K, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Gerber K, Stange G, Roll S, Gauger U, Wiedenmann B, Altenhofen L, Rosch T. Factors determining the quality of screening colonoscopy: a prospective study on adenoma detection rates, from 12,134 examinations (Berlin colonoscopy project 3, BECOP-3). Gut. 2013 Feb;62(2):236-41. doi: 10.1136/gutjnl-2011-300167. Epub 2012 Mar 22. PMID 22442161
- [Background] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301
- [Background] Adler A, Aschenbeck J, Yenerim T, Mayr M, Aminalai A, Drossel R, Schroder A, Scheel M, Wiedenmann B, Rosch T. Narrow-band versus white-light high definition television endoscopic imaging for screening colonoscopy: a prospective randomized trial. Gastroenterology. 2009 Feb;136(2):410-6.e1; quiz 715. doi: 10.1053/j.gastro.2008.10.022. Epub 2008 Oct 15. PMID 19014944
- [Background] Adler A, Pohl H, Papanikolaou IS, Abou-Rebyeh H, Schachschal G, Veltzke-Schlieker W, Khalifa AC, Setka E, Koch M, Wiedenmann B, Rosch T. A prospective randomised study on narrow-band imaging versus conventional colonoscopy for adenoma detection: does narrow-band imaging induce a learning effect? Gut. 2008 Jan;57(1):59-64. doi: 10.1136/gut.2007.123539. Epub 2007 Aug 6. PMID 17681999
- [Background] Adler A, Roll S, Marowski B, Drossel R, Rehs HU, Willich SN, Riese J, Wiedenmann B, Rosch T; Berlin Private-Practice Gastroenterology Working Group. Appropriateness of colonoscopy in the era of colorectal cancer screening: a prospective, multicenter study in a private-practice setting (Berlin Colonoscopy Project 1, BECOP 1). Dis Colon Rectum. 2007 Oct;50(10):1628-38. doi: 10.1007/s10350-007-9029-y. PMID 17694415
- [Background] Pohl H, Aschenbeck J, Drossel R, Schroder A, Mayr M, Koch M, Rothe K, Anders M, Voderholzer W, Hoffmann J, Schulz HJ, Liehr RM, Gottschalk U, Wiedenmann B, Rosch T. Endoscopy in Barrett's oesophagus: adherence to standards and neoplasia detection in the community practice versus hospital setting. J Intern Med. 2008 Oct;264(4):370-8. doi: 10.1111/j.1365-2796.2008.01977.x. Epub 2008 May 15. PMID 18482289
- [Background] Meining A, Ott R, Becker I, Hahn S, Muhlen J, Werner M, Hofler H, Classen M, Heldwein W, Rosch T. The Munich Barrett follow up study: suspicion of Barrett's oesophagus based on either endoscopy or histology only--what is the clinical significance? Gut. 2004 Oct;53(10):1402-7. doi: 10.1136/gut.2003.036822. PMID 15361485
- [Background] Heldwein W, Dollhopf M, Rosch T, Meining A, Schmidtsdorff G, Hasford J, Hermanek P, Burlefinger R, Birkner B, Schmitt W; Munich Gastroenterology Group. The Munich Polypectomy Study (MUPS): prospective analysis of complications and risk factors in 4000 colonic snare polypectomies. Endoscopy. 2005 Nov;37(11):1116-22. doi: 10.1055/s-2005-870512. PMID 16281142
- [Background] Meining A, Driesnack U, Classen M, Rosch T. Management of gastroesophageal reflux disease in primary care: results of a survey in 2 areas in Germany. Z Gastroenterol. 2002 Jan;40(1):15-20. doi: 10.1055/s-2002-19638. PMID 11803496
- [Background] Bajbouj M, Reichenberger J, Neu B, Prinz C, Schmid RM, Rosch T, Meining A. A prospective multicenter clinical and endoscopic follow-up study of patients with gastroesophageal reflux disease. Z Gastroenterol. 2005 Dec;43(12):1303-7. doi: 10.1055/s-2005-858874. PMID 16315125
- [Result] Pioche M, Denis A, Allescher HD, Andrisani G, Costamagna G, Dekker E, Fockens P, Gerges C, Groth S, Kandler J, Lienhart I, Neuhaus H, Petruzziello L, Schachschal G, Tytgat K, Wallner J, Weingart V, Touzet S, Ponchon T, Rosch T. Impact of 2 generational improvements in colonoscopes on adenoma miss rates: results of a prospective randomized multicenter tandem study. Gastrointest Endosc. 2018 Jul;88(1):107-116. doi: 10.1016/j.gie.2018.01.025. Epub 2018 Feb 4. PMID 29410020
- [Result] Zimmermann-Fraedrich K, Groth S, Sehner S, Schubert S, Aschenbeck J, Mayr M, Aminalai A, Schroder A, Bruhn JP, Blaker M, Rosch T, Schachschal G. Effects of two instrument-generation changes on adenoma detection rate during screening colonoscopy: results from a prospective randomized comparative study. Endoscopy. 2018 Sep;50(9):878-885. doi: 10.1055/a-0607-2636. Epub 2018 Jul 23. PMID 30036893